CLINICAL TRIAL: NCT05200143
Title: A Phase II, Single-Arm Clinical Trial Evaluating the Triplet Combination of Ipilimumab, Nivolumab, and Cabozantinib in Patients With Anti-PD-1(L1) Refractory Cutaneous Melanoma
Brief Title: Study of Ipilimumab, Nivolumab, and Cabozantinib in Patients With Cutaneous Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn support from BMS.
Sponsor: Providence Health & Services (Other)
Collaborators: Bristol-Myers Squibb (Industry); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021000533
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Refractory Cutaneous Melanoma
Keywords: Phase 2; Melanoma; ipilimumab; nivolumab; cabozantinib; anti-pd-1
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib + Ipilimumab + Nivolumab (Experimental): Ipilimumab 1 mg/kg + Nivolumab 3 mg/kg IV every 3 weeks + Cabozantinib 40 mg PO daily for 4 cycles followed by Nivolumab 480 mg IV every 4 weeks + Cabozantinib 40 mg PO daily for up to 24 months.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Cabozantinib

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab is a fully human IgG1 kappa monoclonal antibody that binds the co-inhibitory receptor CTLA-4. Antibody binding prevents interaction with the CTLA-4 ligands CD80 and CD86. Blockade of CTLA-4 results in increased T cell activation and proliferation. Ipilimumab was the first immune checkpoint inhibitor to receive FDA approval as a cancer therapy. Treatment of patients with advanced metastatic melanoma with ipilimumab monotherapy resulted in improved overall survival. Subsequent clinical trials with ipilimumab alone and in combination with anti-PD-1 antibodies have demonstrated impressive clinical activity in patients with melanoma, renal cell carcinoma, non-small cell lung cancer and other cancers. Side effects of ipilimumab result from autoimmune attack on healthy tissues. Side effects may include dermatitis, colitis, hepatitis, hypophysitis, pneumonitis, endocrinopathies, nephritis, arthritis, neuropathies and others.
Drug: Nivolumab — Nivolumab is a fully human IgG4 kappa monoclonal antibody that binds the co-inhibitory receptor PD-1. Nivolumab binding to PD-1 blocks interaction with the PD-1 ligands PD-L1 and PD-L2. PD-1 blockade can lead to reinvigoration of exhausted T cells and prevent T cell exhaustion of newly activated T cells. Nivolumab has been shown to have excellent clinical efficacy in treating a wide range of cancers as monotherapy and in combination with ipilimumab.
  Other Names: BMS-936558; MDX1106; ONO-4538
Drug: Cabozantinib — Cabozantinib is a potent small molecule inhibitor of multiple receptor tyrosine kinases. Cabozantinib inhibits VEGFR2, MER, KIT, and MET at single digit nanomolar IC50 concentrations. Other kinases including ROS1, RET, FLT3, RON, AXL, and TIE2 are also inhibited with nanomolar concentrations of cabozantinib. Cabozantinib has been shown to have clinical activity in a variety of solid tumors and has been approved by the FDA for treatment of medullary thyroid cancer, renal cell carcinoma and hepatocellular carcinoma.
  Other Names: XL184

SUMMARY:
The primary objective of this clinical trial is to evaluate the clinical efficacy and progression free survival of the triplet combination of ipilimumab + nivolumab + cabozantinib in patients with anti-PD-1/PD-L1 refractory metastatic cutaneous melanoma.

DETAILED DESCRIPTION:
This is a phase II, single arm, single institution clinical trial. Eligible adults with anti-PD-1 refractory, unresectable/metastatic cutaneous melanoma will be treated with the triplet combination of ipilimumab 1 mg/kg + nivolumab 3 mg/kg every 3 weeks for 4 cycles in addition to cabozantinib 40 mg/day. For cycles 5+, treatment will consist of nivolumab 480 mg IV every 4 weeks in combination with cabozantinib 40 mg/day. The total duration of therapy will be 24 months or until either disease progression or the occurrence of unacceptable drug-related toxicity. Regular tumor assessments should be performed to determine if PD is present.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically (or cytologically) confirmed diagnosis of metastatic cutaneous melanoma.
2. Prior therapy:

   1. Must have been treated previously with an immune checkpoint inhibitor targeting PD-1 or PD-L1.
   2. Disease progression following treatment with prior anti-PD-1/PD-L1 therapy must be confirmed at least 4 weeks after the first imaging showing disease progression to rule out pseudoprogression.
   3. Prior therapy with BRAF/MEK inhibitors (before or after anti-PD-1(L1) therapy) is allowed but not required.
   4. Patients who develop unresectable/metastatic disease while receiving or following completion of adjuvant systemic anti-PD-1/PD-L1 therapy are eligible.
3. Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
4. Men and women, aged ≥ 18 years
5. Measurable disease meeting the following iRECIST criteria:

   1. At least 1 lesion of ≥1.0 cm in the longest diameter for a non-lymph node or >1.5 cm in the short-axis diameter for a lymph node metastasis that is serially measurable according to iRECIST using computed tomography/magnetic resonance imaging (CT/MRI).
   2. Lesions that have had external beam radiotherapy must show evidence of disease progression to qualify as a target lesion.
6. ECOG performance status ≤ 1
7. Adequate cardiac function, as defined by:

   1. Left ventricular ejection fraction (LVEF) ≥ 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram,
   2. Baseline QTc interval ≤ 480 ms
8. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

   1. Absolute neutrophil count (ANC) ≥ 1500/µL without granulocyte colony-stimulating factor support.
   2. White blood cell count ≥ 2500/µL.
   3. Platelets ≥ 100, 000/µL without transfusion.
   4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3x upper limit of normal (ULN). ALP ≤ 5x ULN with documented bone metastases.
   6. Total bilirubin < 1.5 x ULN. Note: Individuals who have a total bilirubin level >1.5 X ULN will be allowed if their indirect bilirubin level is < 1.5 x ULN (i.e., participants with suspected or known diagnosis of Gilbert's Syndrome)
   7. Serum albumin ≥ 2.8 g/dl.
   8. (PT)/INR or partial thromboplastin time (PTT) test < 1.3x the laboratory ULN
   9. Serum creatinine ≤ 1.5x ULN or calculated creatinine clearance ≥ 40mL/min (≥ 0.675mL/sec) using the Cockcroft-Gault equation:

      Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72) Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
   10. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g.
9. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
10. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of cabozantinib and 3 months after the last dose of ipilimumab and 5 months after the last dose of nivolumab.
11. Participants of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at screening, within 24 hours prior to receiving the first dose of study medication, and then every 4 weeks while on treatment.
12. Participants of child-bearing potential agree to use highly effective methods of contraception starting with the first dose of assigned study intervention through 5 months after the last dose of study therapy. Participants of childbearing potential are those who are not proven postmenopausal. Postmenopausal is defined as any of the following:

    1. Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    2. Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
    3. Radiation-induced oophorectomy with last menses >1 year ago
    4. Chemotherapy-induced menopause with >1 year interval since last menses
    5. Surgical sterilisation (bilateral oophorectomy or hysterectomy

Exclusion Criteria:

1. Prior therapy:

   1. Prior systemic therapy within 2 weeks of cycle 1 day 1
   2. Prior therapy with a VEGF(R) inhibitor alone or in combination with immune checkpoint inhibitor(s).
   3. Prior therapy with an anti-CTLA-4 antibody
2. Participants with active, known, or suspected autoimmune disease. Participants with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll.
3. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
4. History of allergy or hypersensitivity to any monoclonal antibody
5. Previous or concurrent malignancy within 3 years of study entry, with the following exceptions:

   1. adequately treated basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy; OR
   2. other solid tumors treated curatively in which the expected rate of recurrence within 5 years is < 5%.
6. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

   1. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) <6 months prior to screening,
   2. Symptomatic congestive heart failure (i.e. Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality <6 months prior to screening. Exceptions include asymptomatic/well-controlled atrial fibrillation/flutter or paroxysmal supraventricular tachycardia;
   3. Uncontrolled hypertension defined as persistent elevation of systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, despite medical therapy
7. History of thromboembolic or cerebrovascular events ≤ 6 months prior to the first dose of study treatment. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e., massive or sub-massive) deep vein thrombosis or pulmonary emboli.

   Note: Individuals with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks.

   Note: Individuals with thromboembolic events related to indwelling catheters or other procedures may be enrolled.
8. Known positive serology for HIV (Human immunodeficiency virus), active hepatitis B, and/or active hepatitis C infection
9. Impaired gastrointestinal function or disease that may significantly alter the absorption of cabozantinib (e.g., uncontrolled vomiting or malabsorption syndrome)
10. Concurrent neuromuscular disorder that is associated with the potential of elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
11. Any other condition that would, in the Investigator's judgment, contraindicate an individual's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
12. Participants who have undergone major surgery (e.g., intracranial, intrathoracic, or intra-abdominal surgery) ≤ 3 weeks prior to starting study drug, minor surgery < 10 days prior to starting study drug or who have not recovered from side effects of such procedure. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment.
13. Participants that are pregnant or nursing (lactating)
14. Prisoners or individuals who are involuntarily incarcerated
15. Medical, psychiatric, cognitive or other conditions that may compromise the participant's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
16. Patients with leptomeningeal involvement by melanoma
17. Participants with CNS metastases or leptomeningeal carcinomatosis are not eligible unless:

    1. CNS metastases have been treated and remained stable by radiographic evaluation at least 4 weeks after CNS directed therapy and/or:
    2. There are ≤5 asymptomatic untreated CNS metastases measuring no larger than 10 mm each.
    3. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment."
18. Radiation therapy for bone metastases within 2 weeks, any other radiation therapy within 4 weeks, or systemic treatment with radionuclides within 6 weeks before first dose of study treatment; ongoing clinically relevant complications from prior radiation therapy are not eligible
19. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:
20. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
21. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
22. Administration of a live, attenuated vaccine within 30 days prior to first dose of study treatment
23. Evidence of tumor invading the GI tract, active peptic ulcer disease, IBD, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of pancreatic duct or common bile duct, or gastric outlet obstruction
24. Abdominal fistula, GI perforation, bowel obstruction or intra-abdominal abscess within 6 months before first dose of study treatment. Complete healing of intra-abdominal abscess must be confirmed before first dose of study treatment
25. Clinically significant hematuria, hematemesis, or hemoptysis of >0.5 tsp (2.5ml) of red blood, or other history of significant bleeding within 12 weeks before first dose of study treatment
26. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
27. Lesions invading or encasing any major blood vessels.
28. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
29. Serious non-healing wound/ulcer/bone fracture.
30. Moderate to severe hepatic impairment (Child-Pugh B or C).
31. Requirement for hemodialysis or peritoneal dialysis.
32. History of solid organ or allogenic stem cell transplant.
33. QTcF > 500 msec within 14 days before first dose of study treatment (Note: Could also be listed in Inclusion as ≤ 500 msec)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Taylor, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was closed early due to withdrawn support from BMS (supplied Nivolumab).
Groups:
- Ipilimumab + Nivolumab + Cabozantinib: Ipilimumab 1 mg/kg + Nivolumab 3 mg/kg IV every 3 weeks + Cabozantinib 40 mg PO daily for 4 cycles followed by Nivolumab 480 mg IV every 4 weeks + Cabozantinib 40 mg PO daily for up to 24 months
Period: Overall Study
Arm/Group | Ipilimumab + Nivolumab + Cabozantinib
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab + Nivolumab + Cabozantinib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) is a measure of functional status from scores ranging from 0 to 5. Baseline measure ECOG PS was collected during the screening physical exam.
  Participants
    ECOG PS 0 (Asymptomatic) | 3
    ECOG PS 1 (Symptomatic but completely ambulatory) | 1
    ECOG PS 2 (Symptomatic, <50% in bed during the day) | 0
    ECOG PS 3 (Symptomatic, >50% in bed, but not bedbound) | 0
    ECOG PS 4 (Bedbound) | 0
    ECOG PS 5 (Death) | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival of the Triplet Combination of Ipilimumab + Nivolumab + Cabozantinib in Patients With Anti-PD-1/PD-L1 Refractory Metastatic Cutaneous Melanoma
Description: Progression free survival (PFS) will be defined as the time between the date of enrollment and the first date of documented progression (per iRECIST), as determined by the investigator, or death due to any cause, whichever occurs first.
Time Frame: 7 Months
Population: 1 of the 4 patients withdrew consent after completing treatment per protocol and moved abroad.
Measure: Median (Full Range); unit: Months
Arm/Group | Ipilimumab + Nivolumab + Cabozantinib
Number analyzed (Participants) | 3
Months | 6.24 [4.60 to 6.37]

2. Secondary Outcome: Safety/Tolerability (CTCAE v5.0)
Description: Number of patients who reported incidence of grade ≥3 treatment related adverse events.
Time Frame: 13 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab + Nivolumab + Cabozantinib
Number analyzed (Participants) | 4
Participants | 2

3. Secondary Outcome: Overall Survival
Description: Number of patients who reached the 12 month overall survival timepoint.
Time Frame: 12 Months
Population: 1 of the 4 patients withdrew consent after completing treatment per protocol and moved abroad.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab + Nivolumab + Cabozantinib
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Description: Adverse events were collected on Day 1 of each cycle. All adverse events collected as part of the study have been reported to ClinicalTrials.gov.
Arm/Group | Ipilimumab + Nivolumab + Cabozantinib
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab + Nivolumab + Cabozantinib (N=4)
Hypophysitis (Endocrine disorders) | 1 (1)
Hepatitis (Infections and infestations) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (2)
Bilateral Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab + Nivolumab + Cabozantinib (N=4)
Abdominal pain/discomfort (Gastrointestinal disorders) | 1 (1)
ALT increased (Investigations) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
AST increased (Investigations) | 2 (5)
Blistering (hands/feet) (Skin and subcutaneous tissue disorders) | 1 (2)
Blood LDH increased (Investigations) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CK increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema, bilateral lower extremity (General disorders) | 1 (1)
Erythematous papular rash, bilateral calves (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Flank pain, right (Musculoskeletal and connective tissue disorders) | 1 (1)
Floaters, intermittent (Eye disorders) | 1 (1)
Hair color changes (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Night Sweats) (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3)
Lipase increased (Investigations) | 1 (2)
Muscle cramp, bilateral feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia, right shoulder/trapezius (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain, right index finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia, bilateral hands/feet (Nervous system disorders) | 1 (1)
Paronychia, intermittent (Infections and infestations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform, scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous papular, chest/abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, bilateral ankles (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (vitiligo) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin pain, palm of left hand (Skin and subcutaneous tissue disorders) | 1 (1)
Skin wound, lower legs (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT05200143/Prot_SAP_001.pdf